CLINICAL TRIAL: NCT03540420
Title: A Randomized Phase II Study Comparing Atezolizumab After Concurrent Chemo-radiotherapy With Chemo-radiotherapy Alone in Limited Disease Small-cell Lung Cancer
Brief Title: Atezolizumab After Concurrent Chemo-radiotherapy Versus Chemo-radiotherapy Alone in Limited Disease Small-cell Lung Cancer
Acronym: ACHILES
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: University Hospital of North Norway (Other); Alesund Hospital (Other); Vestre Viken Hospital Trust (Other); University Hospital, Akershus (Other); Helse Nord-Trøndelag HF (Other); Helse Stavanger HF (Other Government); Haukeland University Hospital (Other); Sorlandet Hospital HF (Other Government); Ullevaal University Hospital (Other); Molde Hospital (Other); Helse Fonna (Other); Nordlandssykehuset HF (Other); Volda Hospital (Other); Kristiansund Hospital (Other); Sahlgrenska University Hospital (Other); Skane University Hospital (Other); Karolinska University Hospital (Other); Ôrebro University Hospital (Unknown); Gävle Hospital (Other); University Hospital, Linkoeping (Other); Odense University Hospital (Other); Aalborg University Hospital (Other); Rigshospitalet, Denmark (Other); National Cancer Center Affiliate of Vilnius University Hospital Santaros Klinikos (Other); Kantonsspital Winterthur KSW (Other); University Hospital, Basel, Switzerland (Other); Insel Gruppe AG, University Hospital Bern (Other); Kantonsspital Graubünden (Other); Freiburger Spital (Other); Klinik Hirslanden, Zurich (Other); Kantonsspital Olten (Other); Spital STS AG (Industry); Ente Ospedaliero Cantonale, Bellinzona (Other); Cantonal Hospital of St. Gallen (Other); St. Olavs Hospital (Other); Oslo University Hospital (Other); Rijnstate Hospital (Other); Isala (Other); Zuyderland Medisch Centrum (Other); The Netherlands Cancer Institute (Other); St. Antonius Hospital (Other); Amphia Hospital (Other); Medisch Spectrum Twente (Other); Erasmus Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-11-03BHG; 2017-004572-62 (EudraCT Number)
Record Dates: First submitted 2018-05-16; First posted 2018-05-30 (Actual); Last update posted 2024-07-15 (Actual); Status verified 2024-07

CONDITIONS: Small-cell Lung Cancer
Keywords: Atezolizumab; Chemoradiotherapy; Immunotherapy
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — atezolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Atezolizumab (Experimental): atezolizumab after completed chemo-radiotherapy and non-progression
  Interventions: Drug: Atezolizumab
- Observation (No Intervention): standard care after completed chemo-radiotherapy and non-progression

INTERVENTIONS:
Drug: Atezolizumab — atezolizumab 1200 mg intravenous every 3 weeks in 12 months
  Other Names: anti-PDL1; Tecentriq
  Arms: Atezolizumab

SUMMARY:
Some patients with limited disease small-cell lung cancer (LD SCLC) are cured after chemo-radiotherapy, but the majority relapse and die from their cancer. Better therapy is needed. Immunotherapy represents the largest advance in cancer therapy in recent years and has demonstrated promising activity in SCLC. In this study we will investigate whether atezolizumab prolongs survival in LD SCLC patients who have undergone chemo-radiotherapy.

DETAILED DESCRIPTION:
Patients who have

* completed 4 course of platinum/etoposide and thoracic radiotherapy of 45 Gy/30 fractions, 2 fractions per day
* non-progression after chemo-radiotherapy
* ECOG performance status 0-2

will be randomized to receive atezolizumab 1200 mg IV every 3 weeks in 12 months or standard of care (observation).

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed small-cell lung cancer
* Previous radiotherapy to the thorax is allowed as long as the patient can receive TRT of 45 Gy.
* Stage I-III according to TNM v8 ineligible for surgery provided all lesions can be included in a tolerable radiotherapy field ("limited disease")
* ECOG performance status 0-2
* Measureable disease according to the RECIST 1.1
* Adequate organ function defined as: (a) Serum alanine transaminase (ALT) ≤ 2.5 x upper limit of normal (ULN); (b) Total serum bilirubin ≤ 1.5 x ULN; (c)Absolute neutrophil count (ANC) ≥ 1.5 x 10 superscr 9/L; (d) Platelets ≥ 100 x 10 superscr 9/L ; (e) Creatinine < 100 µmol/L and calculated creatinine-clearance > 50 ml/min. If calculated creatinine-clearance is < 50 ml/min, an EDTA clearance should be performed
* No malignant cells in pericardial or pleural fluid (at least 1 sample should be obtained if pleural fluid is present) If there is so little fluid that it cannot easily be collected, the patient is considered eligible.
* Pulmonary function: FEV1 > 1 l or > 30 % of predicted value and DLCO > 30 % of predicted value
* Female patients of childbearing potential (Postmenarcheal, not postmenopausal (>12 continuous months of amenorrhea with no identified cause other than menopause), and no surgical sterilization) should use highly effective contraception and take active measures to avoid pregnancy while undergoing atezolizumab treatment and for at least 5 months after the last dose. Birth control methods considered to be highly effective are listed in Appendix D of the protocol
* Written informed consent

Exclusion Criteria:

* previous systemic therapy for SCLC or immune checkpoint blockade therapy
* serious concomitant systemic disorders (for example active infection, unstable cardiovascular disease) which in the opinion of the investigator would compromise the patient's ability to complete the study, or would interfere with the evaluation of the efficacy and safety of the study treatment
* lung disease requiring systemic steroids in doses of >10 mg prednisolone (or equivalent dose of other steroid)
* previous allogeneic or organ transplant
* active or history of autoimmune disease or immune deficiency, including, but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, antiphospholipid antibody syndrome, Wegener granulomatosis, Sjögren syndrome, Guillain-Barré syndrome, or multiple sclerosis
* history of idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis, or evidence of active pneumonitis on screening chest computed tomography (CT) scan
* live vaccine administered in the last 30 days
* active infection requiring IV antibiotics
* active viral hepatitis or HIV-positive
* conditions - medical, social, psychological - which could prevent adequate information and follow-up
* clinically active cancer other than SCLC with the exception of malignancies with a negligible risk of metastases or death (e.g. 5-years OS rate of >90%), such as adequately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma, localized prostate cancer, ductal carcinoma in situ, or stage I uterine cancer. Hormonal therapy for non-metastatic prostate or breast cancer is allowed.
* pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 212 (Actual)
Dates: Start 2018-07-31 (Actual); Primary Completion 2024-04-01 (Actual); Study Completion 2027-04-01 (Estimated)

PRIMARY OUTCOMES:
2 year survival | 2 year after enrollment is completed

SECONDARY OUTCOMES:
Progression free survival | 2 year after enrollment is completed
Best response rate during study treatment period | 2 year after enrollment is completed
Number of treatment-related adverse events as assessed by CTCAE v5.0 | 13 months after last patient completed atezolizumab therapy
  The number of mild (grade 1-2), severe (grade 3-4) and fatal (grade 5) events during the chemoradiotherapy will be reported for the whole study cohort.
Patient-reported Health related quality of life on the EORTC QLQ-C30 and LC13 questionnaires. | 2 year after enrollment is completed
  Patients will report HRQoL before and after chemoradiotherapy and then at each evaluation the first 2 years. Mean scores will be compared at each timepoint. A difference of 10 points or more is considered clinically relevant.

CONTACTS AND LOCATIONS:
Overall Officials: Torstein B Rø, MD, PhD, Study Director — Norwegian University of Science and Technology
Locations (41):
- Denmark (3):
  - Aalborg Universitetshospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Odense University Hospital, Odense
- National Cancer Institute, Vilnius, Lithuania
- Netherlands (8):
  - Antoni van Leeuwenhoek Ziekenhuis, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Amphia Ziekenhuis, Breda
  - Medische Centrum Twente, Enschede
  - Erasmus MC, Rotterdam
  - Zuyderland Ziekenhuis, Sittard
  - Antonius Ziekenhuis, Utrecht
  - Isala Ziekenhuis, Zwolle
- Norway (14):
  - Ålesund Hospital, Ålesund
  - Haukeland Universitetssykehus, Bergen
  - Drammen sykehus - Vestre Viken, Drammen
  - Haugesund hospital, Haugesund
  - Sørlandet Sykehus, Kristiansand
  - Sykehuset i Kristansund, Kristiansund
  - Sykehuset Levanger, Levanger
  - Molde Sjukehus, Molde
  - Akershus Universitetssykehus AHUS, Oslo
  - Oslo University Hospital Ullevål, Oslo
  - Stavanger University Hospital, Stavanger
  - Universitetssykehuset Nord-Norge, Tromsø
  - Cancer Clinic at St. Olavs Hospital, Trondheim
  - Volda hospital, Volda
- Sweden (6):
  - Gävle hospital, Gävle
  - Sahlgrenska Universitetssjukhus, Gothenburg
  - Universitetssjukhuset Linköping, Linköping
  - Skånes University Hospital, Lund
  - Universitetssjukhuset Örebro, Örebro
  - Karolinska University Hospital, Stockholm
- Switzerland (9):
  - Universitätsspital Basel, Basel
  - Inselspital, Bern
  - University Hospital Inselspital, Bern
  - Kantonsspital Graubünden, Chur
  - Kantonsspital Olten - Solothurner Spitäler, Olten
  - Cantonal Hospital of St. Gallen, Sankt Gallen
  - Spital STS AG, Thun
  - Kantonsspital Winterthur, Winterthur
  - Hirslanden Klinik, Zurich

IPD SHARING:
Plan to Share IPD: No